CLINICAL TRIAL: NCT06952777
Title: Measurement and Validation of Fetal Heart and Fetal Movement Signals Detected Via Non-adhesive Sensors
Brief Title: Validation of Sensors for Long-term Non-Invasive Fetal Monitoring
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 107586
Record Dates: First submitted 2025-04-23; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Fetal Distress With Antenatal Problem; Fetal Growth Retardation
Keywords: Fetal monitoring; Fetal heart rate monitoring
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Intervention Model Description: Single arm study comparing sensor output with existing methods of detecting fetal heart rate.
Masking Description: There is no masking of participant or investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women using sensors (Experimental): Participants will be asked to complete a short baseline questionnaire before commencing the monitoring process.
  Participants will be asked to lie on an examination couch for up to 60 minutes at 45 degrees while the electronic sensor(s) are gently held in contact with the maternal abdomen by an elastic belt. In addition to the new sensors the fetal and maternal heart rate will be recorded using the MONICA AN24 device and fetal movements will be recorded with ultrasound (for 20 minutes of the 60). If participants are uncomfortable they will be able to sit or stand to relieve their discomfort.
  Basic information including body mass index, stage of pregnancy and estimated fetal weight will be recorded on a proforma. In addition, participants will be asked to complete a questionnaire about anxiety and wearing the device after the monitoring process.
  Interventions: Other: Non-adhesive capacitively-coupled sensors

INTERVENTIONS:
Other: Non-adhesive capacitively-coupled sensors — Non-adhesive capacitively-coupled sensors which can detect signals of the magnitude of the fetal heart rate and information about fetal movements.

SUMMARY:
A multidisciplinary team of a doctor and engineers have developed a new sensor that will be able to detect mothers' and babies' heartbeat and babies movements in late pregnancy. This sensor can be placed in contact with the mothers' skin over the pregnant uterus without having to be stuck down. We anticipate that this sensor would allow us to monitor babies for longer periods of time which might help us to better identify babies who are being deprived of oxygen during pregnancy. We need to test these sensors on women in late pregnancy for two reasons. Firstly, we need to ensure they reliably measure mother and babies heart rates without interference from movement or other electrical equipment. Secondly we need to ensure that the information they provide is accurate (compared to current measurement techniques).

We will carry out two related studies. The first will include up to 24 women to develop the sensors to ensure that they can obtain consistent signals from mothers' and babies' heartbeats without interference from movement and other electronic devices. We will adjust the electronics in the sensors to ensure they give the best signal. The second will include up to 45 women to see whether the information detected by the sensors is comparable to existing technologies. This information will help us to see whether these sensors can be organised into a new device for fetal monitoring which can then be tested.

DETAILED DESCRIPTION:
In the first part of the study we will ask up to 24 pregnant women to wear the non adhesive sensors and determine whether they consistently detect the electronic signals and to reduce recording of background electrical noise e.g. from electrical wires / devices / sockets etc. which are likely to emit electrical activity in the same microvolt range as the fetal heart rate trace.

Participants will be from three separate time periods in late pregnancy (8 women in each time frame) 28+0-31+6 weeks, 32+0-35+6 weeks and finally from 36+0 until 40+0 weeks. Women will be recruited from the Tommy's research clinics and the antenatal clinics at St Mary's Hospital, Manchester. All participants will have an ultrasound scan prior to participation to measure baby's size, the liquor volume and umbilical artery Doppler (all indicators of baby's wellbeing).

This will ensure that baby is well before the sensors are used. If needed we will make adaptations to the electronics to optimise the detection of the mother's and baby's heart rate.

Participants will be asked to lie on an examination couch for up to 60 minutes at 45 degrees while the electronic sensor(s) are gently held in contact with the maternal abdomen by an elastic belt. If participants are uncomfortable they will be able to sit or stand to relieve their discomfort. Basic information including body mass index, stage of pregnancy and estimated fetal weight will be recorded on a proforma.

If consistent signals can be obtained we will assess whether the sensors can accurately display maternal heart rate and fetal heart rate at different stages of late pregnancy. To assess whether the recording is accurate we will compare the output from the sensors with current methods to assess maternal heart rate (ECG), fetal heart rate (MONICA24).

We will use ultrasound scan to assess whether fetal movements are associated with expected changes in fetal heart activity.

To assess sensor reliability we will recruit up to 15 women from each gestational age group from 28+0-31+6 weeks, 32+0-35+6 weeks and finally from 36+0 until 40+0 weeks. Women will be approached if they have healthy singleton pregnancies and have a pre-pregnancy BMI from 20-35. As previously, women will be recruited from the Tommy's research clinics and the antenatal clinics at St Mary's Hospital, Manchester. The correlation between the maternal and fetal heart rates obtained using established techniques and the new sensors will be calculated.

Participants will be asked to complete a short baseline questionnaire before commencing the monitoring process. Participants will be asked to lie on an examination couch for up to 60 minutes at 45 degrees while the electronic sensor(s) are gently held in contact with the maternal abdomen by an elastic belt. In addition to the new sensors the fetal and maternal heart rate will be recorded using the MONICA AN24 device and fetal movements will be recorded with ultrasound (for 20 minutes of the 60). If participants are uncomfortable they will be able to sit or stand to relieve their discomfort. Basic information including body mass index, stage of pregnancy and estimated fetal weight will be recorded on a proforma. In addition, participants will be asked to complete a questionnaire about anxiety and wearing the device after the monitoring process.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included if they have a non-anomalous singleton pregnancy after 28 weeks' gestation with an estimated fetal weight >10th centile < 90th centile. Participants will be 16 years or over in order that they can give independent consent.

Exclusion Criteria:

* Participants will be excluded if there are fetal anomalies (as defined by the NHS Fetal Anomaly Screening Programme - https://www.gov.uk/guidance/fetal-anomaly-screening-programme-overview), it is a multiple pregnancy, there is evidence of Fetal Growth Restriction (Estimated Fetal Weight <10th centile) or if participants cannot speak or do not understand fluent English. Participants will not be able to participate if they are unable to give informed consent. Participants <16 years of age will be excluded from this study.

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recording quality of non-adherent sensors | 0-60 minutes recording during
  Proportion of recording time that non-adherent sensors record fetal heart rate

SECONDARY OUTCOMES:
Maternal comfort | Immediately after the recording period
  Self-reported comfort of wearing the non-adherent sensors using Likert Scale
Maternal anxiety | Immediately prior to or after the recording period
  Completion of state trait anxiety index

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Heazell, PhD, Principal Investigator — University of Manchester
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data after this initial preclinical study.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT06952777/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT06952777/ICF_001.pdf